CLINICAL TRIAL: NCT03791099
Title: Preparation and Analysis of Material, Biological and Clinical Parameters of Metronidazole-loaded Porous Matrices for Local Periodontitis Treatment
Brief Title: Porous Metronidazole Loaded Matrix for Local Treatment of Periodontitis.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Malgorzata Szulc, Assistant Professor in Periodontology Department, Wroclaw Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB 98/2016
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis treatment; Periodonal pockets; local delivery drugs
MeSH Terms: conditions — Chronic Periodontitis | interventions — Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole (Experimental): 19,8 mg of metronidazole in one polymer matrix
  Interventions: Drug: Metronidazole
- Only SRP (No Intervention): standard non-surgical treatment- scaling/root planing

INTERVENTIONS:
Drug: Metronidazole — After subgingival ultrasonic scaling is performed, metronidazole in polymer matrix is applied to the selected periodontal pockets.
  Arms: Metronidazole

SUMMARY:
Aim of the study is the efficiency assessment of porous Metronidazole loaded matrix based on gelatin/hydroxyethylcellulose blend in treatment of deep periodontal pockets resulting from severe chronic periodontitis. The matrix was invented and produced in Department of Drug Form Technology, Wroclaw Medical University.

The porous metronidazole (MTZ) loaded matrix was fabricated by the freeze-drying technique. The morphology, mechanical properties, in vitro degradation, MTZ release from dried sponge were evaluated and also the clinical trials were performed.

Patients suffering from chronic periodontitis are examined. To evaluate oral hygiene API (Approximal Plaque Index) and the gum inflammation BOP (Bleeding on Probing) and PBI (Papilla Bleeding Index) indices are used. The clinical examination is performed 3 times. On the first visit the output indicators are defined. The subgingival scaling is performed and Metronidazol on porous matrix is applied to the selected periodontal pockets. 2 control tests of periodontal indices are carried out after one week and one month from the application.

In the control group after scaling/root planing procedure, there is no application of metronidazole.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers
* suffering from chronic periodontitis

Exclusion Criteria:

* any antibiotics taken systematically or locally in the preceding six months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
PD | 4 weeks after the first visit
  Periodontal pocket depth
API | 4 weeks after the first visit
  Approximal Plaque Index
BoP | 4 weeks after the first visit
  Bleeding of probing
PBI | 4 weeks after the first visit
  Papilla bleeding index

CONTACTS AND LOCATIONS:
Overall Officials: Marek Ziętek, Prof, Study Chair — Department of Periodontology, Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pandit N, Dahiya R, Gupta R, Bali D, Kathuria A. Comparative evaluation of locally delivered minocycline and metronidazole in the treatment of periodontitis. Contemp Clin Dent. 2013 Jan;4(1):48-53. doi: 10.4103/0976-237X.111615. PMID 23853452
- [Background] Da Rocha HA, Silva CF, Santiago FL, Martins LG, Dias PC, De Magalhaes D. Local Drug Delivery Systems in the Treatment of Periodontitis: A Literature Review. J Int Acad Periodontol. 2015 Jul;17(3):82-90. PMID 26373225
- [Background] Ahmed EM. Hydrogel: Preparation, characterization, and applications: A review. J Adv Res. 2015 Mar;6(2):105-21. doi: 10.1016/j.jare.2013.07.006. Epub 2013 Jul 18. PMID 25750745
- [Background] Gautam S, Dinda AK, Mishra NC. Fabrication and characterization of PCL/gelatin composite nanofibrous scaffold for tissue engineering applications by electrospinning method. Mater Sci Eng C Mater Biol Appl. 2013 Apr 1;33(3):1228-35. doi: 10.1016/j.msec.2012.12.015. Epub 2012 Dec 8. PMID 23827565
- [Background] Pachuau L. Recent developments in novel drug delivery systems for wound healing. Expert Opin Drug Deliv. 2015;12(12):1895-909. doi: 10.1517/17425247.2015.1070143. Epub 2015 Aug 4. PMID 26289672